CLINICAL TRIAL: NCT02590484
Title: The Cervix as a Natural Tamponade in Postpartum Hemorrhage Caused by Placenta Previa and Placenta Previa Accreta: a Prospective Study
Brief Title: The Cervix as a Natural Tamponade in Postpartum Hemorrhage Caused by Placenta Previa and Placenta Previa Accreta
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahmed Rabie Abdelraheim, Dr Ahmed Rabie Abdelraheim, lecturer of Obstetrics And Gynaecology, Minia University
Purpose: Treatment
Other Study IDs: MUH14367
Record Dates: First submitted 2015-10-27; First posted 2015-10-29 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Placenta Previa; Placenta Previa Accreta
MeSH Terms: conditions — Placenta Previa

INTERVENTIONS:
Procedure: The cervix as a natural tamponade (cervical inversion) — Suturing an inverted lip(s) of the cervix over the bleeding placental bed to control the bleeding.
  Other Names: Dawlatly stitch, cervical inversion

SUMMARY:
Placenta previa and placenta accrete carry significant maternal and fetal morbidity and mortality. Several techniques have been described in the literature for controlling massive bleeding associated with placenta previa cesarean sections. The aim of this study is to evaluate the efficacy and safety of the use of the cervix as a natural tamponade in controlling postpartum hemorrhage caused by placenta previa and placenta previa accreta.

DETAILED DESCRIPTION:
Background: Placenta previa and placenta accrete carry significant maternal and fetal morbidity and mortality. The maternal mortality in women with placenta accreta may reach as high as 7-10%. Several techniques have been described in the literature for controlling massive bleeding associated with placenta previa cesarean sections, including uterine packing with gauze, balloon tamponades, the B-Lynch suture, insertion of parallel vertical compression sutures, a square suturing technique and embolization or ligation of the uterine and internal iliac arteries, but there is a wide variation in the success rate of these maneuvers. In a case report, Dawlatly et al. (2007) described a simple technique of suturing an inverted lip of the cervix over the bleeding placental bed that was successful in controlling the bleeding, saving the patient's life, and preserving her uterus.

The objective of this trial is to evaluate the safety and efficacy of the use of this Dawlatly stitch as a natural tamponade for controlling postpartum haemorrhage in cases of placenta previa and/ or placenta previa accreta.

ELIGIBILITY:
Inclusion Criteria:

1. All participating women had one or more previous cesarean deliveries.
2. were diagnosed with placenta previa and/ or placenta previa accreta by ultrasound. When the ultrasound result was not conclusive for placenta accreta, MRI was performed.
3. All participating women desired to preserve their fertility
4. Patients with focal (partial) placenta previa accreta/ placenta previa.

Exclusion Criteria:

1. placenta percreta.
2. diffuse placenta accreta or increta.
3. uncontrollable postpartum hemorrhage.

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Dates: Start 2012-06; Primary Completion 2017-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Successful control of postpartum haemorrhage (PPH) | Intra-operative and up to 24 hours postpartum
  Control of PPH and vaginal bleeding after employing the technique
Number of cases undergoing hysterectomy to control PPH | Intra-operative and up to 24 hours postpartum
  Failure of the technique to stop PPH and need for hysterectomy to stop the bleeding
Incidence of complications | short term (intraoperative and up to 6 weeks postpartum)-long term:up to 2 years postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynaecology, Minia University Hospital, Minya, Egypt

REFERENCES:
- [Derived] El Gelany S, Mosbeh MH, Ibrahim EM, Mohammed M, Khalifa EM, Abdelhakium AK, Yousef AM, Hassan H, Goma K, Alghany AA, Mohammed HF, Azmy AM, Ali WA, Abdelraheim AR. Placenta Accreta Spectrum (PAS) disorders: incidence, risk factors and outcomes of different management strategies in a tertiary referral hospital in Minia, Egypt: a prospective study. BMC Pregnancy Childbirth. 2019 Aug 27;19(1):313. doi: 10.1186/s12884-019-2466-5. PMID 31455286
- [Derived] El Gelany S, Ibrahim EM, Mohammed M, Abdelraheim AR, Khalifa EM, Abdelhakium AK, Yousef AM, Hassan H, Goma K, Khairy M. Management of bleeding from morbidly adherent placenta during elective repeat caesarean section: retrospective -record -based study. BMC Pregnancy Childbirth. 2019 Mar 29;19(1):106. doi: 10.1186/s12884-019-2244-4. PMID 30922265
- [Derived] El Gelany SA, Abdelraheim AR, Mohammed MM, Gad El-Rab MT, Yousef AM, Ibrahim EM, Khalifa EM. The cervix as a natural tamponade in postpartum hemorrhage caused by placenta previa and placenta previa accreta: a prospective study. BMC Pregnancy Childbirth. 2015 Nov 11;15:295. doi: 10.1186/s12884-015-0731-9. PMID 26559634